CLINICAL TRIAL: NCT05676775
Title: British Axial Spondyloarthritis Inception Cohort
Acronym: BAxSIC
Status: Recruiting | Type: Observational
Sponsor: The Leeds Teaching Hospitals NHS Trust (Other)
Responsible Party: Sponsor
Other Study IDs: RR21/146198; 310374 (Other: IRAS)
Record Dates: First submitted 2022-11-24; First posted 2023-01-09 (Actual); Last update posted 2023-07-18 (Actual); Status verified 2023-07

CONDITIONS: Axial Spondyloarthritis
MeSH Terms: conditions — Axial Spondyloarthritis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — HLA-B27 (performed as part of routine clinical care)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: No intervenetion — Observational inception cohort, with remote follow-up via participants and data record linkage

SUMMARY:
The British Axial Spondyloarthritis Cohort (BAxSIC) study has been established under the auspices of the British Society for Spondyloarthritis (BRITSpA) in collaboration with the National Axial Spondyloarthritis Society (NASS) to provide real-world data to evaluate the impact of delay in diagnosis (from symptom onset to diagnosis) on work participation and functional outcomes and the natural history and impact of newly-diagnosed axial Spondyloarthritis, including disease activity, pain, fatigue, functional and work outcomes, comorbidities, therapies in the United Kingdom (UK). The study is a prospective cohort, enrolling patients attending rheumatology clinics in the UK who are newly diagnosed with axial Spondyloarthritis and naïve to biologic therapy.

The study will run for an initial 3 year period commencing January 2023. Financial support was provided as a Research Grant from Pfizer Limited, UCB and Novartis.

DETAILED DESCRIPTION:
Axial spondyloarthritis (axSpA) encompasses a group of chronic rheumatic conditions characterised by inflammation in the axial skeleton. Ankylosing spondylitis (AS) is the prototypic disease, requiring radiographic evidence of sacroiliitis in order to fulfil the modified New York criteria. However, the requirement for radiographic evidence of radiographic sacro-iliac damage in order to make a diagnosis of AS led to long delays (average 10 years) from symptom onset to diagnosis. Furthermore, it was apparent that many patients had symptoms and disability consistent with AS but never developed the required degree of radiographic damage in order to fulfil these criteria. These issues became particularly pressing with the development of effective therapy, initially in the form of TNF (Tumour necrosis factor) inhibitors, for AS. In parallel, advances in magnetic resonance imaging (MRI) enabled the detection of inflammatory changes of sacroiliac joints and the spine prior to the development of structural radiographic damage on plain radiographs. As a result, the Assessment of Spondyloarthritis international Society (ASAS) developed validated classification criteria for axial Spondyloarthritis (axSpA). These criteria allowed a patient chronic back pain to be classified with axSpA via imaging (x-ray or MRI) or clinical (but no imaging) routes, without the requirement for plain film evidence of structural damage. While these classification criteria were initially developed as classification criteria for use in research studies, they have facilitated the earlier diagnosis and treatment of patients with axSpA in clinical practice.

As a result, there have been major advances in AS and axSpA over the past decade. AxSpA has essentially changed from a condition that was diagnosed late, once structural damage was already present, with very limited treatment options to a condition that can now be diagnosed increasingly early and treated with highly effective biologic agents for those with severe disease. There have also been major advances in the understanding of the genetics and pathophysiology of the condition, which has led to the development of new therapeutic agents for SpA, which have already started reaching the clinic years. In combination, these changes have transformed the lives of patients with axSpA.

However, significant unmet need and evidence gaps remain. Studies and audits indicate that despite these advances, there are still delays in diagnosis. The reasons for the delays are likely to be multifactorial but the impact of these delays on outcomes, particularly work and functional, remain poorly defined. This is also compounded by the remaining uncertainty around the natural history of axSpA in real-world settings - only a proportion of people with non-radiographic axSpA (nr-axSpA) will ultimately develop progressive radiographic changes and AS. While other work has started to identify those groups of patients at highest risk of radiographic progression (including those who are HLA-B27 positive, male and/or smokers), accumulating evidence suggests that effective therapy with biologic agents may delay this progression, whilst the long-term impact of early diagnosis and therapy on other outcomes in real-world settings remains unclear. Licensed biologic agents are effective in the management of active axSpA, but remain expensive for health care funders. Thus, longitudinal data are required to help justify their long-term use in real-world settings. Furthermore, despite improvements in inflammation and musculoskeletal symptoms with biologic and non-pharmacological therapies, many people with axSpA have ongoing issues with pain, fatigue, functional and work impairment.

Much of the existing data also comes from clinical trials, which are poorly representative of the general, wider population of people with axSpA. Similarly, clinical trials are usually not of sufficient duration to address long-term impacts of the axSpA spectrum, including extra articular manifestations (EAMs), comorbidities and multimorbidity.

Therefore, there is a requirement for longitudinal, real-world studies of inception cohorts of people diagnosed with axSpA to maximise the benefits from the advances in axSpA, and to address remaining areas of unmet need. This information can also help inform future stratification and precision medicine strategies in axSpA.

ELIGIBILITY:
Inclusion Criteria:

1. Aged ≥16 years.
2. A physician diagnosis of axSpA (including ankylosing spondylitis) within the last 6 months prior to baseline.
3. Willing and able to give informed consent to participate in the study.

Exclusion Criteria:

1. Age <16 years.
2. Unable to communicate in English or are deemed, in any other way, to be unable to give informed consent

Ages: 16 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: The study is a prospective cohort,enrolling patients attending rheumatology clinics in the UK who are newly diagnosed with axial Spondyloarthritis and naïve to biologic therapy.
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2023-06-09 (Actual); Primary Completion 2026-01-09 (Estimated); Study Completion 2029-01-09 (Estimated)

PRIMARY OUTCOMES:
Work Productivity and Activity Impairment (WPAI) | Baseline to 12 months
  Description of baseline characteristics of people with axSpA presenting to rheumatologists and the impact of delay in diagnosis (from symptom onset to diagnosis) on the baseline characteristics at presentation, measured by Work Productivity and Activity Impairment (WPAI).

SECONDARY OUTCOMES:
The Ankylosing Spondylitis Quality of Life index (ASQoL) | 24months
  The Ankylosing Spondylitis Quality of Life index (ASQoL) is a validated disease-specific 18-item questionnaire, that has been developed specifically for measuring health-related quality of life (HRQoL) in subjects with AS. The ASQoL has been used and has shown to be responsive in. The ASQoL score ranges from 0 to 18 with a higher score indicating worse HRQoL.

CONTACTS AND LOCATIONS:
Overall Officials: Helena Marzo-Ortega, MD/PhD, Principal Investigator — Leeds Teaching Hospital Trust
Locations (1):
- Chapel Allerton Hospital, Leeds, United Kingdom

REFERENCES:
- [Derived] Weddell J, Harrison SR, Bennett AN, Gaffney K, Jones GT, Machado PM, Packham J, Sengupta R, Zhao SS, Siebert S, Marzo-Ortega H. British Axial Spondyloarthritis Inception Cohort (BAxSIC): a protocol for a multicentre real-world observational cohort study of early axial spondyloarthritis. Rheumatol Adv Pract. 2024 Jul 26;8(3):rkae087. doi: 10.1093/rap/rkae087. eCollection 2024. PMID 39165398